CLINICAL TRIAL: NCT04281927
Title: A Wearable With Photoplethysmography and 6-lead Electrocardiography for Atrial Fibrillation Detection
Acronym: DoubleCheckAF
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Collaborators: Kaunas University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: S-MIP-17-81
Record Dates: First submitted 2020-01-15; First posted 2020-02-24 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
Keywords: wearable; electrocardiography; photoplethysmography
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atrial fibrillation: Patients with presumed atrial fibrillation will undergo monitoring with the device and Holter ECG.
  Interventions: Device: Monitoring with wearable (the tested device) and Holter ECG (eMotion Faros 90)
- Sinus rhythm: Patients with presumed sinus rhythm will undergo monitoring with the device and Holter ECG.
  Interventions: Device: Monitoring with wearable (the tested device) and Holter ECG (eMotion Faros 90)
- Sinus rhythm and frequent extrasystoles: Patients with presumed sinus rhythm and frequent extrasystoles will undergo monitoring with the device and Holter ECG.
  Interventions: Device: Monitoring with wearable (the tested device) and Holter ECG (eMotion Faros 90)

INTERVENTIONS:
Device: Monitoring with wearable (the tested device) and Holter ECG (eMotion Faros 90) — Participants will use the wearable (the tested device) to record at least 2 minutes of photoplethysmography and 6-lead ECG. In addition, each subject will be monitored with synchronous ECG Holter monitoring (with eMotion Faros 90).

SUMMARY:
A single center prospective case-control study to evaluate ability of a wearable to differentiate between atrial fibrillation (AF) and sinus rhythm (SR).

ELIGIBILITY:
Inclusion Criteria:

* Participants with current ECG-based diagnosis of atrial fibrillation, sinus rhythm or sinus rhythm with frequent (at least once in 2 minutes) premature atrial or ventricular contractions.
* Age is between 18 - 99.

Exclusion Criteria:

* Participants who refuse to sign an informed consent.
* Participants with atrial fibrillation who are currently in a paced rhythm.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of defined groups will be enrolled in Vilnius University Hospital Santaros Clinics.
Sampling Method: Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of a wearable system for atrial fibrillation detection | PPG will be assessed in 2 minutes. ECG will be assessed in up to 10 months.
  The wearable system comprises of two integrated components: a photoplethysmography (PPG) and a 6-lead ECG of the device. It works as described below.
  First, an automatic PPG algorithm will indicate whether atrial fibrillation is suspected. The rhythm assessment of PPG algorithm is based on pulse regularity.
  Next, a 6-lead ECG is acquired by the wearable. The rhythm assessment of ECG is based on P waves and regularity of QRS complexes. A diagnosis is made by independent cardiologists.
  The conclusion of a whole system comprising of both described methods will be compared with a gold standard multi-lead Holter ECG. This standard ECG is also evaluated by independent cardiologists.

SECONDARY OUTCOMES:
Diagnostic accuracy of PPG algorithm of the wearable for atrial fibrillation detection | 2 minutes.
  An automatic PPG algorithm will indicate whether atrial fibrillation is suspected. The rhythm assessment of PPG algorithm is based on pulse regularity. As a separate diagnostic tool it will be compared with a gold standard multi-lead Holter ECG which is assessed by independent cardiologists.
Diagnostic accuracy of a 6-lead ECG of the wearable for atrial fibrillation detection | Up to 10 months.
  Independent cardiologists will assess the heart rhythm in a 6-lead ECG acquired by the wearable. As a separate diagnostic tool it will be compared with a gold standard multi-lead Holter ECG which is also assessed by independent cardiologists. The rhythm evaluation of ECG is based on P waves and regularity of QRS complexes.

CONTACTS AND LOCATIONS:
Overall Officials: Audrius Aidietis, Prof. PhD, Study Chair — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania